CLINICAL TRIAL: NCT01914458
Title: Low-Dose Computed Tomography for Lung Cancer Screening in High Risk Asymptomatic Patients: the Taiwan Study
Brief Title: Image Discovering Early Lung Cancer Project
Acronym: IDEALCAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Cathay General Hosp. IRB, CGHIRB, Cathay General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CGH-LP101004
Record Dates: First submitted 2013-07-28; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Low-dose computed tomography scan
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-dose computed tomography (LDCT) (Experimental): Patients will have one baseline LDCT scan.
  Interventions: Procedure: Low-dose computed tomography (LDCT)

INTERVENTIONS:
Procedure: Low-dose computed tomography (LDCT) — Low-dose computed tomography scan
  Other Names: LDCT scan

SUMMARY:
Lung cancer is the leading cause of cancer related death in Taiwan and world wide. The application of low dose helical computed tomography (CT) has been the milestone of lung cancer screening. Recently, The National Lung Screening Trial (NLST) shows screening with low-dose CT could reduce mortality from lung cancer. We conducted this clinical trial to determine the efficacy of low dose CT in early lung cancer screening in Taiwan.

DETAILED DESCRIPTION:
This is a single center, single arm, non-randomized prospective study. We plan to enroll persons between 50 and 74 years in age, who had cigarette smoking of at least 30 pack-years, and, if former smokers, had quit within the previous 15 years. Persons who had previously received a diagnosis of lung cancer, had undergone chest CT within 18 months before enrollment, had hemoptysis, or had an unexplained weight loss of more than 6.8 kg in the preceding year were excluded.

All the participants should complete a questionnaire that covers many topics, including demographic characteristics and smoking behavior. We also plan to collect additional data for planned analyses of cost-effectiveness, and smoking cessation. Lung-cancer got by biopsy and other biospecimens are available to researchers through a peer-review process All screening examinations are planed to perform in accordance with a standard protocol, developed by medical physicists associated with the trial, that specified acceptable characteristics of the machine and acquisition variables. All low-dose CT scans are acquired with the use of multidetector scanners with a minimum of 16 channels.

IDEALCAP radiologists are certified by appropriate agencies or boards and has completed training in image acquisition; radiologists also has completed training in image quality and standardized image interpretation. Images are interpreted first in isolation and then in comparison with available historical images and images from prior IDEALCAP screening examinations.

IDEALCAP primary analysis is the detection rate of lung cancer. Secondary analysis include the detection rate of lung nodule, 5-year survival rate of persons with lung cancer who receive standard surgical treatment, 5-year survival rate of persons with lung cancer who receive alternative treatment other than standard surgical treatment (ex. Radiotherapy, chemotherapy or target therapy), the correlation of CT images and cigarette smoking history, the correlation of CT images and pulmonary function.

Key Word： low dose computed-tomography (LDCT), lung cancer screening

ELIGIBILITY:
Inclusion Criteria:

* Age 50-74 years
* 30 or more pack-years of cigarette smoking history
* Former smokers: quit smoking within the previous 15 years
* Ability to tolerate CT procedure
* Signed informed consent

Exclusion Criteria:

* Severe uncontrolled heart, vascular, respiratory or endocrine pathology.
* Life-expectancy less than 1 year
* History of lung cancer
* Acute respiratory disease
* Hemoptysis.
* Weight loss more than 6.8 kg in the 12 months prior to eligibility assessment
* Participation in other cancer clinical trial
* Chest CT examination in the 12 months prior to eligibility assessment.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Lung cancer detection rate | 2 years
  Assess number of lung cancer diagnoses after radiological and morphological verification of positive lung nodules.

SECONDARY OUTCOMES:
Lung cancer mortality | 5 years
  Assess lung cancer mortality in the screened group within next 5 years.
All-cause mortality | 5 years
  Assess all-cause mortality mortality within next 5 years.
Nodule detection rate | 3 months
  Estimate nodule detection rate, types (solid, part-solid, or ground glass opacity) and sizes of lung nodules found.
Smoking cessation rate | one year
  Assess smoking cessation rate in the screened group within next one year.

OTHER OUTCOMES:
Coronary artery calcification | 3 months
  Estimate coronary artery calcification score (Agatston Score)in the screened group.
Incidence rate of cardiovascular accident | 5 years
  Incidence rate of cardiovascular accident stratified by coronary artery calcification score in the screened group within next 5 years.
Diagnosis accuracy of COPD diagnosis by low-dose computed tomography(CT) | 2 years
  Assess diagnosis accuracy of COPD diagnosis by low-dose computed tomography(CT) (CT emphysema, CT air trapping) according to the reference standard of pulmonary function tests.
Lung nodules management | 12 months
  Assess algorithms for lung nodules management in a regional general hospital in Taiwan.
Frequency of diagnostic procedures | 12 months
  Estimate the frequency of diagnostic procedures, types of invasive and non-invasive procedures performed in a regional hospital in Taiwan.
Complication of diagnostic procedures | 12 months
  Assess the complication rate after diagnostic procedures performed after screening in a regional hospital in Taiwan. Procedures include baseline LDCT.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Huang Hubert Chan, Doctor, Principal Investigator — CH Chan
Locations (1):
- Lotung Pohai General hospital, Luodong, Taiwan